CLINICAL TRIAL: NCT01910129
Title: A Randomized, Multi-center, Double-blind, Parallel, Crossover Study of a Non-invasive Neurostimulation to the Vagus Nerve With the gammaCore Device for the Reduction in Frequency of Seizures Associated With Epilepsy.
Brief Title: Neurostimulation to the Vagus Nerve for the Reduction in Frequency of Seizures Associated With Epilepsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: E-AU-01; 173/2013 (Other: clinical trail notification)
Record Dates: First submitted 2013-07-15; First posted 2013-07-29 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Seizure
Keywords: vagus nerve stimulation; vagal nerve stimulation; nVNS; VNS; epilepsy; non invasive; gammacore
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gammaCore (Active Comparator): Active stimulation treatment
  Interventions: Device: gammaCore
- sham gammaCore (Placebo Comparator): Inactive stimulation treatment
  Interventions: Device: gammaCore

INTERVENTIONS:
Device: gammaCore — vagal verve stimulation 3 times a day 8 hours apart

SUMMARY:
The purpose of this study is to see the effects of non-invasive vagal nerve stimulation for the reduction in frequency of seizure associated with epilepsy in subjects 18 or older.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of non-invasive vagus nerve stimulation for the reduction in frequency of seizure associated with epilepsy in subjects 18 or older. Subjects will record 4 weeks of baseline seizure activity before being randomized for a period of 8 weeks to receive and active treatment to an active-sham treatment. All subjects will then receive another 8 weeks of active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is diagnosed with epilepsy with; primary generalized tonic-clonic or partial complex or simple complex or focal onset seizures, with or without secondary generalization.
2. The patient's present antiepileptic drug (AED) therapy is ineffective or intolerable
3. The patient is receiving a stable dose of up to 2 oral AED medication(s) and is not expected to have any change in his/her baseline AED treatment during the treatment period.
4. The patient is having more than 2 recordable seizures a month.

Exclusion Criteria:

1. The patient has had status epilepticus within the last six months.
2. The patient has had epilepsy surgery or a VNS implant.
3. The patient has had a history or presence of seizures occurring only in clusters (too frequently or indistinctly separated to be reliably counted).
4. The patient has had 4 weeks continuous seizure freedom last 2 months.
5. The patient has psychogenic non-epileptic seizures (PNES) seizures.
6. The patient has a concomitant progressive CNS disease including progressive myoclonus epilepsy.
7. The patient has a significant history of cardiac, renal, neurologic (other than epilepsy), psychiatric, oncologic, endocrinologic, metabolic, or hepatic disease, which would adversely affect their participation in this study.
8. The patient has had an episode of status epilepticus within 4 weeks of Screening.

10. Has a lesion (including lymphadenopathy), dysaesthesia, previous surgery or abnormal anatomy at the GammaCore treatment site.

11. Has known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g. bruits or history of TIA or CVA), congestive heart failure (CHF), known severe coronary artery disease or recent myocardial infarction.

12. Has an abnormal baseline ECG (e.g. second and third degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction).

13. Has had a previous bilateral, right, or left cervical vagotomy. 14. Has uncontrolled high blood pressure. 15. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.

16. Has a history of carotid endarterectomy or vascular neck surgery on the right side.

17. Has been implanted with metal cervical spine hardware or has a metallic implant near the GammaCore stimulation site.

18. Has a recent or repeated history of syncope. 19. Has a known history or suspicion of substance abuse or addiction. 20. In the opinion of the investigator/research staff the subject is incapable of operating the GammaCore device as intended and performing the data collection procedures.

21. Is pregnant, nursing, thinking of becoming pregnant in the next 9 months, or of childbearing years and is unwilling to use an accepted form of birth control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Beran, Professor, Principal Investigator
Locations (2):
- Australia (2):
  - Southern Neurology, Kogarah, New South Wales
  - Strategic Health Evaluators, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No
The study was prematurely discontinued

RESULTS

PARTICIPANT FLOW:
Groups:
- gammaCore Then Sham gammaCore: 8 weeks active stimulation with the gammaCore device , no wash out , followed by 8 weeks sham treatment with the sham device
  gammaCore/sham treatment: vagal verve stimulation 3 times a day 8 hours apart
- Sham gammaCore Then gammaCore: 8 weeks sham treatment with the sham device, no wash -out, followed by 8 weeks sham treatment with the with the gammaCore device
  gammaCore/sham treatment: vagal verve stimulation 3 times a day 8 hours apart
- Run-in Period: Not randomized or allocated to treatment group
Period: Run-in Period Phase 1
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore | Run-in Period
Started | 0 | 0 | 13
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 0
Period: Randomized Phase 2
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore | Run-in Period
Started | 7 | 6 | 0
Completed | 5 | 5 | 0
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Period: Randomized Phase 3
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore | Run-in Period
Started | 5 | 5 | 0
Completed | 5 | 4 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- gammaCore Then Sham gammaCore: 8 weeks Active gammaCore stimulation treatment followed by 8 weeks sham (inactive) gammaCore treatment
  gammaCore: vagal verve stimulation 3 times a day 8 hours apart
- Sham gammaCore Then gammaCore: 8 weeks sham (inactive) gammaCore treatment followed by 8 weeks active gammaCore treatment
  gammaCore: vagal verve stimulation 3 times a day 8 hours apart
- Total: Total of all reporting groups
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Full Range); unit: years] | 43 [23 to 66] | 59 [46 to 68] | 51 [23 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 4 | 10
  Asian | 0 | 2 | 2
  Indian (Fiji) | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Seizures
Description: The seizure frequency was collected in the subject diary throughout Intervention 1/Phase 2 (8 weeks) and Intervention 2/Phase 3 (8 weeks).
Time Frame: 16 weeks
Population: safety population 3 subjects were missing data in phase 3 (2 from phase 2 active group and 1 from the phase 2 sham group)
Measure: Mean (Full Range); unit: seizures
Groups:
- gammaCore Then Sham gammaCore: Active gammaCore stimulation treatment followed by sham gammaCore treatment
  gammaCore: vagal verve stimulation 3 times a day 8 hours apart
- Sham gammaCore the gammaCore: Inactive sham gammaCore stimulation treatment followed by Active gammaCore stimulation
  gammaCore: vagal verve stimulation 3 times a day 8 hours apart
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore the gammaCore
Number analyzed (Participants) | 7 | 6
seizures
  Frequency of Seizure Phase 2 | 9.1 [2 to 17] | 8.2 [2 to 21]
  Frequency of Seizure Phase 3: number analyzed (Participants) | 5 | 5
  Frequency of Seizure Phase 3 | 9.4 [2 to 17] | 6.6 [0 to 12]

2. Secondary Outcome: Duration of Seizure
Description: Duration of seizure was recorded by the subject in the subject diary throughout Intervention 1/Phase 2 (8 weeks) and Intervention 2/Phase 3 (8 weeks).
Time Frame: 16 weeks
Population: Safety population. One subject has missing data in the active gammacore group. 2 subjects were missing data in phase 3 (1 from phase 2 active group and 1 from the phase 2 sham group)
  1 subject in the phase 3 sham group reported 0 seizures during this phase
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- gammaCore Then Sham gammaCore: Active gammaCore stimulation treatment followed by inactive sham gammaCore treatment
  gammaCore: vagal verve stimulation 3 times a day 8 hours apart
- Sham gammaCore Then gammaCore: Inactive sham gammaCore stimulation treatment followed by active gammaCore treatment
  gammaCore: vagal verve stimulation 3 times a day 8 hours apart
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore
Number analyzed (Participants) | 6 | 6
minutes
  Duration of Seizure Phase 2 | 4.5 (4.3) | 6.5 (10.7)
  Duration of Seizure Phase 3: number analyzed (Participants) | 5 | 4
  Duration of Seizure Phase 3 | 6.0 (8.5) | 5.9 (7.2)

3. Secondary Outcome: Severity of Seizure
Description: The Seizure Severity Questionnaire (SSQ) is a self-reported assessment tool, which categorizes seizures into three phases: warning, ictal activity and postictal recovery. The recovery phase is subdivided into three components (cognitive, emotional and physical aspects of recovery), each of which is rated for frequency, severity and bothersome. Overall assessment of seizure severity is measured with the last two items.
  Items are positively scored from a scale of 1-7, with lower scores representing a better status. 1 = none, never or mild and 7 = extremely frequent, severe or high.
  The severity was reported for seizures occuring throughout Intervention 1/Phase 2 (8 weeks) and Intervention 2/Phase 3 (8 weeks).
Time Frame: 16 weeks
Population: Safety population. 4 subjects were missing data (one in the gammacore group and 3 in the sham group) 3 subjects in the gammacore group were missing data in phase 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore
Number analyzed (Participants) | 6 | 3
units on a scale
  Severity of Seizure Phase 2 | 4.0 (2.14) | 2.8 (2.24)
  Severity of Seizure Phase 3: number analyzed (Participants) | 3 | 3
  Severity of Seizure Phase 3 | 4.8 (2.70) | 4.0 (1.49)

4. Secondary Outcome: Type of Adverse Events
Description: Type of adverse events were split in to Adverse Events, Adverse Device Effects and Serious Adverse Events. Adverse events were reported throughout Intervention 1/Phase 2 (8 weeks) and Intervention 2/Phase 3 (8 weeks).
  For frequency see the Adverse Event Table.
Time Frame: 16 weeks
Population: Safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Run-in Phase 1: No treatment - 4 week run-in phase
- gammaCore Phase 2; gammaCore Phase 3: gammaCore stimulation treatment
  gammaCore: vagal verve stimulation 3 times a day 8 hours apart
- Sham Phase 2; Sham Phase 3: sham gammaCore stimulation treatment
  sham stimulation 3 times a day 8 hours apart
Arm/Group | Run-in Phase 1 | gammaCore Phase 2 | Sham Phase 2 | gammaCore Phase 3 | Sham Phase 3
Number analyzed (Participants) | 13 | 7 | 6 | 5 | 5
Participants
  Adverse Device Effect | 0 | 5 | 4 | 2 | 2
  Adverse Events | 6 | 5 | 4 | 2 | 4
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Seizure Free Days
Description: The number of seizure-free days was collected from the subjects' diary. The total number of days observed days for each phase and the total number of seizure free days for each phase are presented for the course of the study throughout Intervention 1/Phase 2 (8 weeks) and Intervention 2/Phase 3 (8 weeks).
Time Frame: 16 weeks
Population: Safety population. 1 subject was missing data in the gammacore group.
  1 subject from phase 2 gammacore group and 1 subject from the phase 2 sham group were missing data in phase 3
Measure: Number; unit: days
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore
Number analyzed (Participants) | 6 | 6
days
  Phase 2 Number of observed days (total) | 295 | 281
  Phase 2 Number of observed seizure free days | 257 | 245
  Phase 3 Number of observed days (total): number analyzed (Participants) | 5 | 5
  Phase 3 Number of observed days (total) | 296 | 270
  Phase 3 Number of observed seizure free days: number analyzed (Participants) | 5 | 5
  Phase 3 Number of observed seizure free days | 255 | 244

6. Secondary Outcome: Quality of Life in Epilepsy
Description: The Quality of Life in Epilepsy-31 (QOLIE-31) instrument is a self- administered questionnaire. It includes seven subscales: Overall Quality of Life, Seizure Worry, Emotional Well-Being, Energy/Fatigue, Cognitive, Medication Effects, and Social Function. Questions 1-30 can yield seven individual scores (per subtest) and a total (composite) score. Higher scores indicate better QOL with values ranging from 1 to 100.
  Question 31 is a subjective assessment of one's general health condition.Higher scores indicate a better-reported general health condition with the range being 1-10.
  Scores are presented at end of Intervention 1/Phase 2 (8 weeks) and at the end of Intervention 2/Phase 3 (8 weeks).
Time Frame: 16 weeks
Population: Safety population. 2 subject in the gammacore group and 1 subject in the sham group were missing data.
  1 subject in the gammacore group was missing data in phase 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | gammaCore Then Sham gammaCore | Sham gammaCore Then gammaCore
Number analyzed (Participants) | 5 | 5
units on a scale
  Phase 2 Questions 1-30 | 55 (11.72) | 63 (19.74)
  Phase 2 Question 31 | 7 (1.48) | 6 (1.95)
  Phase 3 Questions 1-30: number analyzed (Participants) | 4 | 5
  Phase 3 Questions 1-30 | 55 (24.61) | 59 (17.95)
  Phase 3 Question 31: number analyzed (Participants) | 4 | 5
  Phase 3 Question 31 | 7 (2.78) | 6 (2.19)

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- Run-in Phase 1: Not randomized or allocated to treatment group
- gammaCore Phase 2; gammaCore Phase 3: 8 weeks gammaCore stimulation treatment
  gammaCore vagal verve stimulation 3 times a day 8 hours apart
- Sham Phase 2; Sham Phase 3: 8 weeks sham stimulation treatment
  sham stimulation 3 times a day 8 hours apart
Arm/Group | Run-in Phase 1 | gammaCore Phase 2 | Sham Phase 2 | gammaCore Phase 3 | Sham Phase 3
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7 | 0/6 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 6/13 | 5/7 | 4/6 | 2/5 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase 1 (N=13) | gammaCore Phase 2 (N=7) | Sham Phase 2 (N=6) | gammaCore Phase 3 (N=5) | Sham Phase 3 (N=5)
Increased seizure frequency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in left leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in left shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pains in left ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Period pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right hand pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain left anterior chest wall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Broken sleep (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drowsy (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Unusual feeling in nose (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Unusual feeling in the mouth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nose tingle right side (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash in left ear (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling of withdrawal from medication (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tired eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Change of appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prominent veins (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epiphora (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red spot/bite on both legs (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling of indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feel bloated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Difficulty concentrating (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pinched nerve (back) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left forearm injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right ankle pinched nerve (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low blood pressure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Light headed, dizzy, slight nausea, double vision (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shoulder ache arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor in both hands (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scab on neck (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
tennis elbow returned (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Damaged sciatic nerve (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right eustachian tube blockage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 2 (5) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of balance (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired hearing right ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bland taste (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort at site of stimulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Paresthesia on top and bottom lip on right side during treatment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia at site of stimulation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling funny - face and arms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metal taste in mouth during treatment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Paresthesia in neck and underarms (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parethesia teeth (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vagus nerve stimulation feels abrasive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fillings irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching at site of stimulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle pain at site of stimulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash on neck (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dull pain on right side of neck going up to right side of head (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less